CLINICAL TRIAL: NCT04656392
Title: Early Detection of Barrett's Esophagus and Esophageal Cancer: Accuracy and Acceptability of a Novel Screening Strategy in Primary Care
Brief Title: Early Detection of Barrett's Esophagus in Participants With Reflux Symptoms in Primary Care
Acronym: ELECTRONIC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Collaborators: Dutch Digestive Diseases Foundation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 110769
Record Dates: First submitted 2020-11-30; First posted 2020-12-07 (Actual); Last update posted 2024-04-16 (Actual); Status verified 2024-04

CONDITIONS: Barrett Esophagus; Esophageal Cancer
Keywords: Barrett Esophagus; Esophageal Cancer; Primary care; General practice; Screening
MeSH Terms: conditions — Barrett Esophagus; Esophageal Neoplasms | interventions — Breath Tests

STUDY DESIGN:
Intervention Model Description: The study design is a multi-site prospective cohort study in eight general practices. All participants will receive the breath test with the eNose in the general practice, followed by the uTNE in the hospital.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Breath test (eNose) followed by uTNE. (Other): All participants will receive the breath test with the eNose in the general practice, followed by the uTNE in the hospital.
  Interventions: Diagnostic Test: Breath test (eNose) followed by uTNE.

INTERVENTIONS:
Diagnostic Test: Breath test (eNose) followed by uTNE. — All participants will receive the breath test with the eNose in the general practice, followed by the uTNE in the hospital.

SUMMARY:
In the Netherlands, the incidence of esophageal adenocarcinoma (EAC) is increasing. In addition, EAC has a dismal prognosis. Therefore, screening for Barrett's Esophagus (BE) has stimulated interest. Although BE is a known precursor of EAC, a minority of patients with EAC are known with a previous diagnosis of BE. A non-invasive screening tool, such as breath testing, could select patients at risk for BE, after which unsedated transnasal endoscopy (uTNE) can confirm or exclude the diagnosis. The objective is to determine the accuracy and acceptability of a non-invasive screening strategy i.e. breath testing followed by uTNE for BE and EAC.

DETAILED DESCRIPTION:
The ongoing increasing incidence of esophageal adenocarcinoma (EAC) in the Netherlands during the last few decades and the still dismal prognosis has stimulated interest in screening for Barrett's esophagus (BE). Although BE is a known precursor of EAC, a minority of patients with EAC (<10%) are known with a previous diagnosis of BE, and hence, most cases of BE are undiagnosed. Screening programs to detect BE followed by endoscopic surveillance and treatment of dysplasia or early neoplasia seem able to reduce the incidence of EAC and improve survival. A non-invasive screening tool, such as breath testing, could select patients at risk for BE, after which unsedated transnasal endoscopy (uTNE) can confirm or exclude the diagnosis. uTNE offers the possibility of a more acceptable and accurate endoscopic assessment of the esophagus with almost neglectable risks and lower costs compared to conventional endoscopy. The objective is to determine the accuracy and acceptability of a non-invasive screening strategy i.e. breath testing followed by uTNE for BE and EAC.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged 50 to 75 years;
* Recorded diagnosis of reflux symptoms >90 days OR
* Recorded prescriptions for acid suppressant therapy for this indication for at least 1 year in the past 5 years
* Written informed consent.

Exclusion Criteria:

* Upper endoscopy in the previous 5 years;
* A current or previous diagnosis and/or treatment of any type of malignancy (not including basal-cell skin cancer (BCC) and squamous-cell skin cancer (SCC)) within the last five years;
* Already known with a diagnosis of Barrett's esophagus or gastro-esophageal cancer;
* Any argument provided by a patient's own general practitioner not to include the patient;
* Comorbidities precluding transnasal endoscopy (e.g. inability to discontinue oral anticoagulants, history of recurrent epistaxis, allergy to lidocaine derivatives).

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 449 (Actual)
Dates: Start 2021-04-20 (Actual); Primary Completion 2024-03-11 (Actual); Study Completion 2024-03-11 (Actual)

PRIMARY OUTCOMES:
Positive Predictive Value (PPV) of the eNose for detecting confirmed BE | 16 weeks after breath test (eNose)
  PPV of the eNose for detecting confirmed BE with the diagnosis made by transnasal endoscopy and upper endoscopy as the reference standard in primary care.
Negative Predictive Value (NPV) of the eNose for detecting confirmed BE | 16 weeks after breath test (eNose)
  NPV of the eNose for detecting confirmed BE with the diagnosis made by transnasal endoscopy and upper endoscopy as the reference standard in primary care.
Sensitivity of the eNose for detecting confirmed BE | 16 weeks after breath test (eNose)
  Sensitivity of the eNose for detecting confirmed BE with the diagnosis made by transnasal endoscopy and upper endoscopy as the reference standard in primary care.
Specificity of the eNose for detecting confirmed BE | 16 weeks after breath test (eNose)
  Specificity of the eNose for detecting confirmed BE with the diagnosis made by transnasal endoscopy and upper endoscopy as the reference standard in primary care.

SECONDARY OUTCOMES:
Patient acceptability (discomfort and overall experience) of the eNose measured on a NPRS. | Directly after breath test (eNose)
  Patient acceptability consists of two questions regarding discomfort and overall experience of the eNose. Discomfort is measured on a Numeric Pain Rating Scale (NPRS) with 0 being 'none' and 10 being 'severe'. Overall experience is measured on a Numeric Pain Rating Scale (NPRS) with 0 being 'the worst experience', 5 being 'neither pleasant nor unpleasant' and 10 being 'the best experience'.
Patient acceptability (discomfort and overall experience) of uTNE measured on a NPRS. | Directly after uTNE
  Patient acceptability consists of two questions regarding discomfort and overall experience of uTNE. Discomfort is measured on a Numeric Pain Rating Scale (NPRS) with 0 being 'none' and 10 being 'severe'. Overall experience is measured on a Numeric Pain Rating Scale (NPRS) with 0 being 'the worst experience', 5 being 'neither pleasant nor unpleasant' and 10 being 'the best experience'.
Patient acceptability (discomfort and overall experience) of conventional endoscopy (if applicable) measured on a NPRS. | Directly after conventional endoscopy
  Patient acceptability consists of two questions regarding discomfort and overall experience of conventional endoscopy. Discomfort is measured on a Numeric Pain Rating Scale (NPRS) with 0 being 'none' and 10 being 'severe'. Overall experience is measured on a Numeric Pain Rating Scale (NPRS) with 0 being 'the worst experience', 5 being 'neither pleasant nor unpleasant' and 10 being 'the best experience'.
Willingness to undergo repeat eNose procedure | Directly after breath test (eNose)
  Willingness to undergo repeat procedure consists of one question with answer options 'Yes' and 'No'.
Willingness to undergo repeat uTNE procedure | Directly after uTNE
  Willingness to undergo repeat procedure consists of one question with answer options 'Yes' and 'No'.
Willingness to undergo repeat conventional endoscopy | Directly after conventional endoscopy
  Willingness to undergo repeat procedure consists of one question with answer options 'Yes' and 'No'.
Cancer worry (CWS-8) | At baseline, 7 days after eNose, 7 days after uTNE, 7 days after conventional endoscopy (if applicable), 30 days after eNose, 30 days after uTNE, 30 days after conventional endoscopy (if applicable), 90 days after last study procedure.
  The Cancer Worry Scale (CWS-8) is used to measure cancer worry. Scores are ranging from 8 to 32, and higher scores indicate more cancer worry.
Anxiety (STAI-6) | At baseline, 7 days after eNose, 7 days after uTNE, 7 days after conventional endoscopy (if applicable), 30 days after eNose, 30 days after uTNE, 30 days after conventional endoscopy (if applicable), 90 days after last study procedure.
  The State-Trait Anxiety Inventory (STAI-6) is used to measure anxiety. Scores are ranging from 6 to 24, and higher scores indicate more anxiety.
Impact of event (IES-15) | 7 days after eNose, 7 days after uTNE, 7 days after conventional endoscopy (if applicable), 30 days after eNose, 30 days after uTNE, 30 days after conventional endoscopy (if applicable), 90 days after last study procedure.
  The Impact of Event Scale (IES-15) is used to measure impact of event. Scores are ranging from 0 to 75, and higher scores indicate more impact of event.
Rate of successful evaluation by uTNE | 1 week after the last participant undergoes uTNE.
  The rate of successful intubation and complete evaluation will be measured.
Rate of successful evaluation by breath test (eNose) | 1 week after the last participant undergoes breath test (eNose).
  The rate of successful intubation and complete evaluation will be measured.
Safety of uTNE based on reported Adverse Events. | 1 week after the last participant undergoes uTNE.
  The safety will be measured based on reported Adverse Events.
Safety of eNose based on reported Adverse Events. | 1 week after the last participant undergoes breath test (eNose).
  The safety will be measured based on reported Adverse Events.

CONTACTS AND LOCATIONS:
Overall Officials: Peter D. Siersema, Prof.dr., Principal Investigator — Radboud University Medical Center Nijmegen
Locations (1):
- Radboud University Medical Center, Nijmegen, Gelderland, Netherlands

IPD SHARING:
Plan to Share IPD: No